CLINICAL TRIAL: NCT02612545
Title: A Multi-Site, Open-Label, Randomized Trial to Assess the Efficacy, Safety, and Tolerability of Dihydroartemisinin-Piperaquine Plus Mefloquine Compared to Dihydroartemisinin-Piperaquine or Artesunate-Mefloquine in Patients With Uncomplicated Falciparum Malaria in Cambodia
Brief Title: Efficacy, Safety, and Tolerability of Dihydroartemisinin-piperaquine + Mefloquine Compared to Dihydroartemisinin-piperaquine or Artesunate-mefloquine in Patients With Uncomplicated Falciparum Malaria in Cambodia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999916023; 16-I-N023
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10-08

CONDITIONS: Acute Falciparum Malaria
Keywords: Plasmodium Falciparum; Artemisinin Combination Therapy; Triple Artemisinin Combination Therapy; Piperaquine; Mefloquine
MeSH Terms: conditions — Malaria, Falciparum | interventions — Mefloquine

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (2):
- ACT (Active Comparator): Patients randomized to ACT will receive DHA-PPQ only
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHA-PPQ)
- TACT (Experimental): Patients randomized to TACT will receive DHA-PPQ plus MQ
  Interventions: Drug: Dihydroartemisinin-piperaquine (DHA-PPQ); Drug: Mefloquine (MQ)

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine (DHA-PPQ) — Co-formulated anti-malarial drug used as standard of care treatment for uncomplicated malaria in Cambodia
Drug: Mefloquine (MQ) — ACT partner drug
  Arms: TACT

SUMMARY:
Background:

Malaria is an illness caused by a parasite that enters people s bodies when a mosquito bites them. It can cause fevers, headaches, body aches, and weakness. If not treated, it can make some people very ill. Malaria can be cured. A mix of 2 drugs that has worked well in the past is not working as well in some parts of Cambodia. Researchers want to see if a mix of 3 drugs works better and is safe.

Objectives:

To see if a 3-drug mix can be used to treat malaria in areas where a 2-drug mix is less effective.

Eligibility:

People aged 2 65 years with mild malaria in Pursat, Preah Vihear, and Ratanakiri Provinces in Cambodia.

Design:

Participants will be screened with medical history, physical exam, urine and blood tests, and an electrocardiogram (ECG). For this, electrodes will be placed on their skin to check their heartbeat.

Participants will spend about 5 nights in the hospital. They will have physical exams and will complete symptom questionnaires daily. They will give blood periodically throughout their stay. For this, a thin plastic tube is placed in an arm vein for the first day, and blood draws using a needle are done after that.

Participants will get either a 2-drug mix or a 3-drug mix for 3 days. They will have 2 ECGs each day of receiving the drugs.

Participants will have follow-up visits once a week over 5 weeks. At these visits, they will have a physical exam and have blood taken. If they have any signs of malaria, they will be re-treated.

The study will last up to 42 days.

DETAILED DESCRIPTION:
Dihydroartemisinin-piperaquine (DHA-PPQ) Cambodia s frontline artemisinin (ART) combination therapy (ACT) for Plasmodium falciparum malaria is failing to cure nearly half of patients in its western provinces. These treatment failures are caused by parasite strains that are resistant to both ART and PPQ, yet sensitive to mefloquine (MQ) in vitro and in vivo. These findings, and previous studies showing that PPQ treats MQ-resistant infections in patients, led us to hypothesize that parasites have not developed cross-resistance to both PPQ and MQ. Given that DHA-PPQ and AS+MQ have both failed rapidly to resistance when used alone, we propose to treat patients with triple ACT (TACT) containing DHA-PPQ + MQ. We believe that this TACT will more effectively cure patients than either ACT alone, and will continue to achieve acceptably high cure rates and help to eliminate malaria in Cambodia until new drugs are developed and deployed. This protocol thus aims to measure the efficacy, safety, and tolerability of DHA-PPQ + MQ versus DHA-PPQ or AS-MQ alone in a multi-site, open-label, randomized clinical trial. In each of three Cambodian provinces (Pursat, Preah Vihear, and Ratanakiri) where DHA-PPQ is failing, we will recruit subjects aged 2 to 65 years with uncomplicated falciparum malaria (randomized 1:1), In Pursat and Preah Vihear we will treat them with either DHA-PPQ + MQ or AS-MQ alone and in Ratanakiri we will treat them with either DHA-PPQ + MQ or DHA-PPQ alone for three days, and follow them for 42 days to assess for recrudescent parasitemia an indicator of treatment failure. The main safety concern of this study is that DHA-PPQ + MQ may cause electrocardiographic (ECG) changes that could predispose a patient to develop clinically significant arrhythmias. This is because PPQ is known to cause prolongation of the ECG corrected QT (QTc) interval, and MQ may further increase PPQ levels (and thus the risk of further QTc prolongation) through pharmacokinetic interactions involving CYP3A4, a liver enzyme that metabolizes both drugs. To monitor for such an event, we will obtain ECG recordings before and after each drug dose. The safety and tolerability of TACT versus ACT will also be assessed through periodic tests of hematopoietic, hepatic, and renal function, and frequent symptom questionnaires. We will also administer a single low dose of primaquine, which kills P. falciparum gametocytes, on Day 2 to interrupt the transmission of parasites to mosquitoes and promote the elimination of malaria in Cambodia. During hospitalization and followup, we will obtain a series of research blood samples to estimate the prevalence of genetic markers for ART, PPQ, and MQ resistance; to develop a genotyping platform for rapidly surveying known drug resistance-associated mutations; investigate the genomic and transcriptomic basis of drug-resistance mechanisms; confirm the elimination of parasites and gametocytes from the bloodstream using sensitive molecular methods; measure the ex-vivo susceptibility of parasites to antimalarial drugs, and cryopreserve parasites for future studies to elucidate the molecular mechanisms of drug resistance.

ELIGIBILITY:
* INCLUSION:
* Age 2 to 65 years
* Uncomplicated falciparum malaria, confirmed by the presence of asexual P.falciparum parasites (alone or mixed with other Plasmodium species) on blood film
* Asexual P. falciparum count <200,000/ L at screening
* Tympanic temperature greater than or equal to 37.5 (Infinite)C or history of fever in the previous 24 hours
* Written informed consent from adults or the parents/guardians of children

EXCLUSION:

* Signs of severe malaria, defined as one or more of the following:
* Glasgow Coma Scale less than or equal to 10/15 in adults; Blantyre Coma Scale less than or equal to 3/5 in children

  * Witnessed convulsions
  * Severe prostration
  * Shock (poor perfusion, cool peripheries as deemed by the study physician)
  * Hematocrit <20%
  * Jaundice
  * Respiratory distress (labored breathing, nasal flaring, intercostal retraction)
  * Anuria for 24 hours or more
  * Repetitive vomiting
* Hematocrit <25%
* Acute illness other than uncomplicated falciparum malaria requiring treatment
* Pregnancy or breastfeeding
* Patients who have received an ART derivative or ACT in the previous 7 days
* Treatment with MQ in the previous 60 days
* History of allergy or known contraindication to ART, PPQ, MQ, or PMQ
* Splenectomy
* Documented or claimed history of cardiac arrythmias, neuropsychiatric disease
* Earlier participation in this trial
* Any condition that in the opinion of the investigator would render the patient unable to comply with the protocol (e.g., psychiatric disease)
* Any health condition that in the opinion of the investigator would confound data analysis (e.g., patients known to be HIV-infected or to have AIDS) or pose unnecessary exposure risks to the patient (e.g., severe malnutrition)

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2015-11-20; Primary Completion 2018-10-12 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of TACT versus ACT, as defined by an adequate clinical and parasitological response (ACPR), defined as: absence of parasitemia on Day 42 (detected by blood smear, not PCR), irrespective of tympanic temperature, in subjects w... | Day 42 post enrollment

SECONDARY OUTCOMES:
Compare parasite and fever clearance rates/times following TACT versus ACT | Days 0-6 post enrollment
Compare the safety and tolerability of TACT versus ACT | Day 0-6 post enrollment
Compare ECG QTc prolongation following TACT versus ACT | Days 0-2 post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Wellems, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Center for Parasitology, Entomology, and Malaria Controk, Ministry of H, Phnom Penh, Cambodia

REFERENCES:
- [Background] Ashley EA, Dhorda M, Fairhurst RM, Amaratunga C, Lim P, Suon S, Sreng S, Anderson JM, Mao S, Sam B, Sopha C, Chuor CM, Nguon C, Sovannaroth S, Pukrittayakamee S, Jittamala P, Chotivanich K, Chutasmit K, Suchatsoonthorn C, Runcharoen R, Hien TT, Thuy-Nhien NT, Thanh NV, Phu NH, Htut Y, Han KT, Aye KH, Mokuolu OA, Olaosebikan RR, Folaranmi OO, Mayxay M, Khanthavong M, Hongvanthong B, Newton PN, Onyamboko MA, Fanello CI, Tshefu AK, Mishra N, Valecha N, Phyo AP, Nosten F, Yi P, Tripura R, Borrmann S, Bashraheil M, Peshu J, Faiz MA, Ghose A, Hossain MA, Samad R, Rahman MR, Hasan MM, Islam A, Miotto O, Amato R, MacInnis B, Stalker J, Kwiatkowski DP, Bozdech Z, Jeeyapant A, Cheah PY, Sakulthaew T, Chalk J, Intharabut B, Silamut K, Lee SJ, Vihokhern B, Kunasol C, Imwong M, Tarning J, Taylor WJ, Yeung S, Woodrow CJ, Flegg JA, Das D, Smith J, Venkatesan M, Plowe CV, Stepniewska K, Guerin PJ, Dondorp AM, Day NP, White NJ; Tracking Resistance to Artemisinin Collaboration (TRAC). Spread of artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2014 Jul 31;371(5):411-23. doi: 10.1056/NEJMoa1314981. PMID 25075834
- [Background] Leang R, Taylor WR, Bouth DM, Song L, Tarning J, Char MC, Kim S, Witkowski B, Duru V, Domergue A, Khim N, Ringwald P, Menard D. Evidence of Plasmodium falciparum Malaria Multidrug Resistance to Artemisinin and Piperaquine in Western Cambodia: Dihydroartemisinin-Piperaquine Open-Label Multicenter Clinical Assessment. Antimicrob Agents Chemother. 2015 Aug;59(8):4719-26. doi: 10.1128/AAC.00835-15. Epub 2015 May 26. PMID 26014949
- [Background] Spring MD, Lin JT, Manning JE, Vanachayangkul P, Somethy S, Bun R, Se Y, Chann S, Ittiverakul M, Sia-ngam P, Kuntawunginn W, Arsanok M, Buathong N, Chaorattanakawee S, Gosi P, Ta-aksorn W, Chanarat N, Sundrakes S, Kong N, Heng TK, Nou S, Teja-isavadharm P, Pichyangkul S, Phann ST, Balasubramanian S, Juliano JJ, Meshnick SR, Chour CM, Prom S, Lanteri CA, Lon C, Saunders DL. Dihydroartemisinin-piperaquine failure associated with a triple mutant including kelch13 C580Y in Cambodia: an observational cohort study. Lancet Infect Dis. 2015 Jun;15(6):683-91. doi: 10.1016/S1473-3099(15)70049-6. Epub 2015 Apr 12. PMID 25877962